CLINICAL TRIAL: NCT01357564
Title: Nonpharmacologic Management of Challenging Behaviors in Veterans With Dementia
Brief Title: Tailored Activity Program-Veterans Affairs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IIR 11-119
Record Dates: First submitted 2011-05-18; First posted 2011-05-20 (Estimated); Results first posted 2019-03-22 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2018-12

CONDITIONS: Dementia
Keywords: dementia; caregivers; tailored activity; neuropsychiatric symptoms; behavioral symptoms
MeSH Terms: conditions — Dementia; Behavioral Symptoms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tailored Activity Program (Experimental): Occupational therapists assess the person's home environment, preserved capabilities, daily routines, interests and the caregiver's readiness and ability to use activities. Activities are developed that reflect the Veteran's previous or current interests and are modified to match their preserved capabilities without taxing the most impaired areas of cognition (e.g., memory, new learning). TAP-VA provides caregivers with the knowledge and skills to use activities. The overall goal is to provide predictability, familiarity, and structure in the daily life of the Veteran and establish a level of environmental stimulation appropriate to that person's abilities.
  Interventions: Other: Tailored Activity Program
- Attention Control (Active Comparator): Caregivers in this group receive bi-weekly telephone contact by a trained healthcare professional. In each session, caregivers are provided important information about dementia and strategies for disease management. Each telephone contact begins with a brief overview of the specific purpose of the session, followed by a description of the key facts about the session topic, and concludes with a question and answer period. The attention control group intervention is delivered by a member of the research team who is knowledgeable about dementia and has had prior experience working with family caregivers.
  Interventions: Other: Attention Control

INTERVENTIONS:
Other: Tailored Activity Program — The interventionist, an occupational therapist, meets with the caregiver and introduces the intervention goals. The OT provides and reviews written educational materials about dementia, importance of taking care of self, communication strategies and other educational materials. Also provided and reviewed is The 36 Hour Day. The OT interviews the caregiver to obtain information about previous roles, habits, past and current daily routines, caregiver and Veteran preferences and interests. The OT also observes interactions, noting communication and management style. The OT will also meet with the Veteran, observe social capacity using the Peavy Comportment scale and administer the Dementia Rating Scale.
  Arms: Tailored Activity Program
Other: Attention Control — Caregivers in this group received bi-weekly telephone contact by a trained healthcare professional. In each session, caregivers were provided information about dementia and strategies for disease management. Each telephone contact began with a brief overview the session purpose, followed by a description of key facts, and concluded with a question and answer period. The attention control group intervention was delivered by a member of the research team who is knowledgeable about dementia and has had prior experience working with family caregivers.
  Arms: Attention Control

SUMMARY:
The Tailored Activity Program - Veterans Administration is a Phase III efficacy trial designed to reduce behavioral symptoms in Veterans with dementia living with their caregivers in the community. The study uses a randomized two group parallel design with 160 diverse Veterans and caregivers. The experimental group receives a transformative patient-centric intervention designed to reduce the burden of behavioral symptoms in Veterans with dementia. An occupational therapist conducts an assessment to identify a Veteran's preserved capabilities, deficit areas, previous roles, habits, and interests to develop activities tailored to the Veteran. Family caregivers are then trained to incorporate activities into daily care. The attention-control group receives bi-monthly telephone contact where education on topics relevant to dementia is provided to caregivers. Key outcomes include reduced frequency and severity of behavioral symptoms using the 12-item Neuropsychiatric Inventory (primary endpoint), reduced caregiver burden, enhanced skill acquisition, efficacy using activities, and time spent providing care at 4 months; and long-term effects (8 months) on the Veteran's quality of life and frequency and severity of behavioral symptoms, and caregiver use of activities. The programs' impact of Veterans Administration cost is also examined. Study precision will be increased through face-to-face research team trainings with procedural manuals and review of audio-taped interviews and intervention sessions.

DETAILED DESCRIPTION:
This study tests the efficacy of a transformative patient-centric intervention designed to reduce the burden of NPS in Veterans with dementia who live at home with family caregivers. The innovative intervention, the Tailored Activity Program (TAP-VA), involves 8 sessions over 4 months in Veterans' homes. An occupational therapist conducts a systematic assessment to identify a Veteran's preserved capabilities and deficit areas, and previous roles, habits and interests from which to develop and introduce activities tailored to the Veteran's profile. Family caregivers are then trained to incorporate tailored activities into daily care routines. The intervention was pilot tested in an NIMH funded study with 60 community-living individuals with dementia. Findings from this pilot showed statistically significant and clinically meaningful reductions in NPS, specifically agitation and less time being on "duty" by family caregivers. Results of this pilot phase support moving forward with a full-scale Phase III efficacy trial. The investigators tested TAP-VA in a randomized two-group parallel design in which 160 racially and ethnically diverse Veterans with dementia and their family caregivers (dyads) were randomly assigned to receive TAP-VA or an attention control group. All dyads were evaluated at baseline and 4-months (main trial endpoint), and then reassessed at 8-months to evaluate long-term treatment effects (baseline to 8 months), including continued activity use, caregiver well-being, and costs.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Veterans with dementia include:

* English speaking
* diagnosed with dementia as above
* able to participate in at least two activities of daily living

  * ADLs - bathing
  * dressing
  * grooming
  * toileting
  * transferring from bed to chair
* not currently participating in any other dementia-related intervention.
* If the Veteran with dementia is on any of four classes of psychotropic medications:

  * antidepressant
  * benzodiazepines
  * antipsychotic
  * anti-convulsant
  * an anti-dementia medication (memantine or a cholinesterase inhibitor)
* We will require that he/she have been on a stable dose for 60 days prior to enrollment to minimize possible confounding effects of concomitant medications (the typical time frame used in clinical trials).
* Caregivers of Veterans must be:

  * English speaking
  * self-identify as the primary member of the family caring (hands-on or supervision) for the Veteran and 21 years of age or older (male or female)
  * living with the Veteran
  * accessible by telephone to schedule interview, intervention sessions and follow-up interviews
  * planning to live in area for 8 months (to reduce loss to follow-up)
  * indicate willingness to learn activity use
  * report one or more NPS in the Veteran in the past month
  * not currently participating in any other caregiver-related intervention.
* Finally, we will require that caregivers taking a psychotropic medication (antidepressant, benzodiazepines, antipsychotic, or anti-convulsant) at time of telephone screen be on a stable dose of the medication for 60 days prior to enrollment.

Exclusion Criteria:

* Non English speaking
* Non-Veteran
* No caregiver
* No diagnosis of dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2012-08; Primary Completion 2016-06 (Actual); Study Completion 2018-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ivette Freytes, PhD MS BS, Principal Investigator — North Florida/South Georgia Veterans Health System, Gainesville, FL
Locations (1):
- North Florida/South Georgia Veterans Health System, Gainesville, FL, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gitlin LN, Mann WC, Vogel WB, Arthur PB. A non-pharmacologic approach to address challenging behaviors of Veterans with dementia: description of the tailored activity program-VA randomized trial. BMC Geriatr. 2013 Sep 23;13:96. doi: 10.1186/1471-2318-13-96. PMID 24060106
- [Result] Gitlin LN, Arthur P, Piersol C, Hessels V, Wu SS, Dai Y, Mann WC. Targeting Behavioral Symptoms and Functional Decline in Dementia: A Randomized Clinical Trial. J Am Geriatr Soc. 2018 Feb;66(2):339-345. doi: 10.1111/jgs.15194. Epub 2017 Nov 28. PMID 29192967
- See also: Alzheimer's information site — http://www.alz.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Tailored Activity Program: Intervention Group
  Tailored Activity Program: Intervention Protocol: In session #1, the interventionist, an occupational therapist (OT), meets with the caregiver and introduces the intervention goals. The OT provides and reviews a 3-ring binder which contains written educational materials about dementia, importance of taking care of self, communication strategies and other educational materials. Also provided and reviewed will be a copy of Mace and Rabins' book, The 36 Hour Day. The OT will interview the caregiver to obtain information about previous roles, habits, past and current daily routines, caregiver and Veteran preferences and interests. The OT will also observe interactions, noting communication and management style. The OT will also meet with the Veteran, observe social capacity using the Peavy Comportment scale and administer the Dementia Rating Scale (DRS-2).
- Attention Control: Attention Control
Period: Short-term (4-month) Follow up
Arm/Group | Tailored Activity Program | Attention Control
Started | 154 | 168
Completed | 106 | 118
Not Completed | 48 | 50
Period: Long-term (8-month) Follow-up
Arm/Group | Tailored Activity Program | Attention Control
Started | 106 | 118
Completed | 104 | 102
Not Completed | 2 | 16

BASELINE CHARACTERISTICS:
Groups:
- Tailored Activity Program: Tailored intervention activity.
  Tailored Activity Program: Intervention Protocol: In session #1, the interventionist, an occupational therapist (OT), meets with the caregiver and introduces the intervention goals. The OT provides and reviews a 3-ring binder which contains written educational materials about dementia, importance of taking care of self, communication strategies and other educational materials. Also provided and reviewed will be a copy of Mace and Rabins' book, The 36 Hour Day. The OT will interview the caregiver to obtain information about previous roles, habits, past and current daily routines, caregiver and Veteran preferences and interests. The OT will also observe interactions, noting communication and management style.
- Attention Control: Attention control.
  Caregivers in this group receive bi-weekly telephone contact (up to 8 contacts) by a trained healthcare professional. In each session, caregivers are provided important information about dementia and strategies for managing the disease at home (Table 2). Each telephone contact is approximately 30 minutes in length and begins with a brief overview of the specific purpose of the session, followed by a description of the key facts about the session topic, and concludes with a question and answer period. Table 2 outlines the specific domain and session content that is covered. The attention control group intervention is delivered by a member of the research team who is knowledgeable about dementia and has had prior experience working with family caregivers.
- Total: Total of all reporting groups
Arm/Group | Tailored Activity Program | Attention Control | Total
Number analyzed (Participants) | 154 | 168 | 322
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 28 | 52
  >=65 years | 130 | 140 | 270
Age, Continuous [Mean (Full Range); unit: years] | 77.43 [33 to 100] | 71.34 [47 to 91] | 76.21 [33 to 100]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 84 | 161
  Male | 77 | 84 | 161
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 6
  Not Hispanic or Latino | 150 | 165 | 315
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 20 | 33 | 53
  White | 129 | 127 | 256
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 8 | 13
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 154 | 168 | 322

OUTCOME MEASURES:

1. Primary Outcome: The Neuropsychiatric Inventory (NPI). Measures the Frequency and Severity of Behavioral Symptoms in Dementia.
Description: The Neuropsychiatric Inventory (NPI) assesses the frequency and severity of 12 common behavioral symptoms in dementia.
  The NPI Score is calculated by multiplying the total reported frequency by the severity score, with a theoretical range of 0-1704: high scores indicating greater frequency by severity.
  The change between 2 or more time points is being reported. Baseline to T2 (4 months) - short-term measure; and baseline to T3 (8 months) - long term measure
Time Frame: Baseline, 4 month (short-term follow-up), 8 month (long-term)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Tailored Activity Program: The INT is designed to draw on residual abilities of Veterans with dementia and provide an environment supportive of these abilities. Occupational therapists assess the person's home environment, preserved capabilities, daily routines, interests and the caregiver's readiness and ability to use activities. Activities are developed that reflect the Veteran's previous or current interests and are modified to match their preserved capabilities without taxing the most impaired areas of cognition (e.g., memory, new learning). TAP-VA provides caregivers with the requisite knowledge and skills to use activities. Caregivers are instructed in specific skills such as ways to simplify activities, the environment and their communication, and how to help the Veteran initiate and follow a sequence. The overall goal is to provide predictability, familiarity, and structure in the daily life of the Veteran and establish a level of environmental stimulation appropriate to that person's abilities.
- Attention Control: The ATN Serves 3 purposes: 1) creates clinical equipoise, ensuring that ethical treatment is provided to all study participants; 2) controls for the one-on-one attention to caregivers in the intervention group to rule out potential effects of professional contact; and 3) serves as a retention tool. Caregivers in this group receive bi-weekly telephone contact by a trained healthcare professional. In each session, caregivers are provided important information about dementia and strategies for disease management. Each telephone contact begins with a brief overview of the specific purpose of the session, followed by a description of the key facts about the session topic, and concludes with a question and answer period. Table 2 outlines the specific domain and session content that is covered. The attention control group intervention is delivered by a member of the research team who is knowledgeable about dementia and has had prior experience working with family caregivers.
Arm/Group | Tailored Activity Program | Attention Control
Number analyzed (Participants) | 154 | 168
score on a scale
  T1-T2 (sort term) Change | -38.1 [-50.33 to -25.86] | 1.0 [-11.8 to 13.8]
  T1-T3 (long term) Change | -12 [-23.22 to -0.78] | -9.8 [-20.19 to .58]
Statistical Analysis 1: Comparison: Tailored Activity Program vs Attention Control; Sample size calculation was based on the main study hypothesis tested at 80% power for a 2-sided alternative hypothesis using a t-test comparing the treatment groups on 4-month values. Based on previous trials, we sought a medium effect size of 0.50 using a type I error rate of .05; Test type: Superiority; p = .02, t-test, 2 sided; Mean Difference (Net) = -.72, 95% CI 2-sided [-1.23 to -0.13]

2. Secondary Outcome: 12-item Zarit Burden Short Form Measuring Caregiver Burden
Description: Caregiver burden as measured by the 12-item Zarit Burden Short Form.
  Scores range from 0-48, with higher scores indicating burden; scores over 17 indicate particularly high levels of caregiver burden.
  The change between 2 or more time points is being reported. Baseline to T2 (4 months) - short-term measure; and baseline to T3 (8 months) - long term measure
Time Frame: Baseline, 4 month (short-term follow-up), 8 month (long-term)
Measure: Number; unit: units on a scale
Groups:
- Tailored Activity Intervention: Tailored Activity Program: Intervention
- Attention Control: Phone calls/education
Arm/Group | Tailored Activity Intervention | Attention Control
Number analyzed (Participants) | 154 | 168
units on a scale
  T1-T2 (short term) change | -1.4 | -1.6
  T1-T3 (long term) change | -0.7 | 0.01
Statistical Analysis 1: Comparison: Tailored Activity Intervention vs Attention Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .03, t-test, 2 sided; Mean Difference (Net) = -.1, 95% CI 2-sided [-0.14 to -0.01]

ADVERSE EVENTS:
Arm/Group | Tailored Activity Program | Attention Control
All-Cause Mortality (participants affected / at risk) | 5/154 | 9/168
Serious Adverse Events (participants affected / at risk) | 7/154 | 4/168
Other Adverse Events (participants affected / at risk) | 0/154 | 0/168
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tailored Activity Program (N=154) | Attention Control (N=168)
Hospitalization/Rehab (Congenital, familial and genetic disorders) | 7 (7) | 4 (4)

LIMITATIONS AND CAVEATS:
Study limitations include use of a single veteran setting, small sample size, and that medication change effects are unclear.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2014-11-17): https://cdn.clinicaltrials.gov/large-docs/64/NCT01357564/Prot_000.pdf